CLINICAL TRIAL: NCT06775158
Title: Perioperative Myocardial and Renal Injury in Patients Undergoing Hepatic Resection: Incidence, Risk Factors, Predictors and Relation with Patient Outcomes: a Retrospective Cohort Study
Brief Title: Perioperative Myocardial and Renal Injury in Patients Undergoing Hepatic Resection
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Specialist in Anesthesiology and Reanimation, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 27..2024.297
Record Dates: First submitted 2025-01-04; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Liver Neoplasm; Kidney Injury, Acute; Myocardial Injury After Non-Cardiac Surgery
Keywords: Hepatic resection; acute kidney injury; perioperative myocardial injury
MeSH Terms: conditions — Liver Neoplasms; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with organ injury: Patitents who suffered from AKI or PMI
- Patients without organ injury: Patitents who did not suffer from AKI or PMI

SUMMARY:
Liver surgeries are high risk surgeries that might result in injuries in kidneys and heart. This study was planned to investigate the frequency of these injuries as well as the risk factors for their devolopment and its effect on patient outcomes.

DETAILED DESCRIPTION:
Hepatic resections are highly invasive major surgical procedures and are associated with higher incidence of end-organ injuries, specifically acute kidney injury (AKI) and perioperative myocardial injury (PMI). This study was designed to determine the incidences of AKI and PMI, and reveal the risk factors for their development and investigate intraoperative labaratory predictors in patients undergoing hepatic resection. We also planned to evaluate the relationship between the occurrence of end-organ injury and length of hospital and intensive care unit (ICU) stay, and 90-day mortality.

Patients were identified from a prospectively maintained data file that involves the perioperative data of patients undergoing surgery at Hepatobiliary-Pancreas clinic of Başakşehir Çam&Sakura City Hospital. All consequtive patients within the study period were evaluated for inclusion. 128 patients were eligible for statistical analysis. This sample size was sufficient to determine the incidence of perioperative organ injury with a margin error of 8.4%. Green formula revealed that the sample size was sufficient for evaluating 9 variables in a regression model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hepatic resection

Exclusion Criteria:

* presence of end stage kidney disease
* emergency surgery
* application of total vascular exclusion
* concomitant gastrointestinal resection
* duration of surgery less than 100 minutes
* non-oncologic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent resection in Hepatobiliary&Pancreatic Surgery Clinic of Başakşehir Çam&Sakura City Hospital, between june 2021 and june 2024
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients sufferd from Acute Kidney injury | 3 days postoperatively
  at least 0.3mg/dL or 50% increase from baseline creatinine levels within 3 days postoperatively is described as Acute Kidney İnjury. Data will be presented as frequency(percentage) and the margin error of the percentage
Number of patients suffered from Perioperative myocardial injury | 3 days postoperatively
  At least 14 ng/L increase from baseline high sensitive Troponin T levels within 3 days psotoperatively is described as perioperative myocardial injury. Data will be presented as frequency(percentage) and the margin error of the percentage
Number of patients suffered from perioperative organ injury | 3 days postoperatively
  Occurence of acute kidney injury or perioperative myocardial injury within 3 days in patients undergoing hepatic resection. Descriptions are clarified in the prior outcomes' description sections. Data will be presented as frequency(percentage) and the margin error of the percentage
Odds Ratios of Risk Factors for the Occurence of perioperartive organ injury | 3 days postoperatively
  Patients' demographic, medical and intraoperative characteristics will be evaluated in terms of the occurence of perioperative organ injury. Variables with the p value < 0,05 will be added to the logistic regression model.

SECONDARY OUTCOMES:
Length of intensive care unit stay | 90 days postoperatively
  Length of intensive care unit stay during postoperative period will be evaluated in patients who did and did not suffer from perioperative organ injury
Length of hospital stay | 90 days postoperatively
  Length of hospital stay in the postoperative period, including intensive care will be evaluated in patients who did and did not suffer from perioperative organ injury
90-day mortality | 90 days postoperatively
  90-day mortality following the surgery will be evaluated in patients who did and did not suffer from perioperative organ injury

OTHER OUTCOMES:
Area under the curve of receiver operating characteristics curve generated by using intraoperative Lactate, base excess, venous saturation and delta carbondioxide pressure | 3 days postoperatively
  intraoperative labaratory parameters obtained by arterai blood gas analysis will be evaluated by creating a model with logistic regression

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam&Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All raw data that will be used during the statitistical analysis will be shared by the primary investigator upon reosanable request